CLINICAL TRIAL: NCT04264702
Title: BESPOKE Study of ctDNA Guided Therapy in Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Natera, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 20-041-NCP
Record Dates: First submitted 2020-02-04; First posted 2020-02-11 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Colorectal Cancer; Colon Cancer
Keywords: circulating tumor DNA; BESPOKE
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — There are two arms to this study: A prospective arm that will enroll 2000 patients, and a historical control (retrospective arm) that will enroll 600 patients.
  Each participant in the Prospective arm will have received the commercially available SIGNATERA™ test.
  Subjects prospectively enrolled and whom consent to "Optional future Research" may have bio-specimens stored for future research. The historical arm (retrospective cohort) will not have any bio-specimens collected or stored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective arm: Patients who have undergone surgery for stage I to IV colorectal cancer (CRC) and who have residual formalin-fixed paraffin-embedded (FFPE) tissue available will provide FFPE and whole blood samples. Patients will receive SIGNATERA™ test results and may be recommended for adjuvant chemotherapy or observation by their treating clinician. Patients will be followed for up to two years with periodic whole blood collection. Treatment administered, disease-free survival, overall survival, time to recurrence, physician questionnaires and patient-reported outcomes will be recorded.
- Control Arm: The control arm will consist of matched Stage I to Stage IV CRC cases using the following criteria: sex, age of diagnosis and ECOG performance prior to ACT, and a minimum of 3 evaluations per year. The patient cases would have a minimum of 2 years follow-up data and received treatment no more than 3 years prior to study start date.

SUMMARY:
The BESPOKE CRC study will prospectively enroll patients who have undergone surgery for stage I to IV colorectal cancer (CRC) and who have residual formalin-fixed paraffin-embedded (FFPE) tissue available will provide FFPE and whole blood samples. Patients will receive SIGNATERA™ test results and may be recommended for post-operative systemic therapy or observation by their treating clinician. Patients will be followed for up to two years with periodic whole blood collection. The study also has a control arm that will consist of matched Stage I to IV CRC cases that have a minimum of least 2 years clinical follow-up data.

DETAILED DESCRIPTION:
Primary Objectives:

* Examine the impact of SIGNATERA™ on adjuvant treatment decisions
* Determine the rate of recurrence of patients diagnosed with CRC while asymptomatic using SIGNATERA™

Secondary objectives:

* Molecular residual disease clearance as assessed by SIGNATERA™
* Percent of patients undergoing surgery for oligometastatic recurrence
* Survival in patients treated with adjuvant versus no adjuvant chemotherapy in patients with SIGNATERA™ negative test results
* Overall survival
* Impact of SIGNATERA™ test results on patient quality of life

ELIGIBILITY:
Inclusion criteria:

1. 18 years of age or older.
2. Planning or undergone surgical resection of adenocarcinoma of the colon or rectum.
3. Diagnosis of Colorectal cancer that falls into one of the below categories:

   1. Stage I to IV disease.
   2. Stage IV with oligometastatic disease eligible for post-operative systemic therapy.
4. Selected by their healthcare provider to receive the SIGNATERA™ test according to the current evidence-informed schedule as part of their routine practice.
5. ECOG performance status ≤ 2
6. Clinically eligible for post-operative systemic therapy.
7. Able to tolerate venipuncture for research blood draw(s).
8. Able to read, understand and provide written informed consent .
9. Willing and able to comply with the study requirements.

Exclusion Criteria:

1. Pregnant or breastfeeding.
2. Prior history and treatment for any cancer within the past year or has another active cancer, with the exception of non-melanoma skin cancer
3. Has a known rare inherited genetic condition, with the exception of lynch syndrome
4. Has initiated post-operative systemic therapy.
5. Neuropathy > grade 2.
6. History of bone marrow or organ transplant.
7. Medical condition that would place the patient at risk as a result of blood donation, such as bleeding disorder .
8. Serious medical condition that may adversely affect ability to participate in the study.

Control Arm Inclusion criteria:

1. 18 years of age or older at time of diagnosis.
2. Diagnosis of Colorectal cancer that falls into one of the below categories:

   1. Stage I to IV disease.
   2. Stage IV with oligometastatic disease eligible for post-operative systemic therapy.
3. Were clinically eligible for chemotherapy at full recommended doses per Health Care Provider.
4. Received treatment no more than 3 years prior to study start date.
5. Have a minimum of least 2 years clinical follow-up data or reached a progression event.

Control Arm Exclusion criteria:

1. Female patients that were pregnant or breastfeeding during historical control collection period.
2. Per investigator, was not clinically eligible for post-operative systemic therapy.
3. Had an ECOG performance status ≤ 2 at time of diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been diagnosed with Stage I, Stage II, Stage III or Stage IV colorectal cancer.
Sampling Method: Probability Sample
Enrollment: 1788 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Examine the impact of SIGNATERA™ on adjuvant treatment decisions | 1 years
  The study will examine the percent of patients who have their adjuvant treatment regimen increased or decreased after the treating physician evaluates the results from the post-surgical SIGNATERA™ ctDNA test for patients with Stage II and Stage III CRC.
Determine the rate of recurrence of patients diagnosed with CRC while asymptomatic using SIGNATERA™ | 2 years
  The study will examine the Proportion of positive SIGNATERA™ results at any timepoint during surveillance; prior to being identified by other methods whilst undergoing recurrence monitoring for patients with Stage I to IV CRC

SECONDARY OUTCOMES:
Evaluate Molecular residual disease clearance as assessed by SIGNATERA™ | 2 years
  The proportion of patients with a positive SIGNATERA™ ctDNA test post-surgery that subsequently receive a negative test result during or after systemic therapy
The study will examine the percent of patients undergoing surgery for oligometastatic recurrence | 2 years
  The proportion of patients that are diagnosed with oligometastatic recurrence that undergo additional surgery
Evaluate survival in patients treated with adjuvant versus no adjuvant chemotherapy in patients with SIGNATERA™ negative test results | 2 years
  Proportion of patients with a negative SIGNATERA™ ctDNA test post-surgery that are still alive the end of the trial (during surveillance) treated with adjuvant versus no adjuvant chemotherapy
Explore Overall survival | 2 years
  Proportion of patients with a negative SIGNATERA™ ctDNA that are still alive the end of the trial (during surveillance)
Examine the Impact of SIGNATERA™ test results on patient quality of life | 2 years
  Determine if SIGNATERA™ results makes patients feel less worried or anxious about the possibility of cancer recurrence. Assess if SIGNATERA™ makes patients feel that they are receiving the right treatment and determine if patients would continue to use Signatera in the future to monitor their cancer recurrence. This will be measured by asking the patients three study specific questions on a 5-point scale (1=Not all, 5= All the time) with a lower score indicating a better outcome.
Assess well being in patients receiving SIGNATERA™ ctDNA test results | 2 years
  Assess a patients wellbeing using the National Comprehensive Cancer Network Functional Assessment of Cancer Therapy Colorectal Symptom Index- 19 items (NCCN-FACT FCIS-19 version 2). Responses for each items are given on a 4-point scale (0=Not at all, 4 = very much) with a lower score indicating a better outcome.
Assess patient cancer anxiety levels in patients receiving SIGNATERA™ ctDNA test results | 2 years
  Assess Fear of Recurrence in patients receiving SIGNATERA™ ctDNA test results by using the Fear of Recurrence short form (FCR-4) using a 5-point scale (1=Not all, 5= All the time) with a lower score indicating a better outcome.
Assess patient anxiety and depression levels in patients receiving SIGNATERA™ ctDNA test results | 2 years
  Assess patient anxiety and depression levels in patients receiving SIGNATERA™ ctDNA test results using the Hospital Anxiety and Depression Scale (HADS-A). The HADS is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. The anxiety and depression subscales each range from 0 to 21, with higher scores indicating higher anxiety/depression complains. Patients were defined as having anxiety or depression or both if the score was 8 or more in the corresponding subscale.
Examine the number of Stage I CRC patients that have recurrent disease detected post-surgery based on SIGNATERA™ test results | 2 years
  Proportion of Stage I CRC cases with a positive SIGNATERA™ test and have recurrent disease detected post-surgery and receive systemic therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Aleshin, MD, MBA, Principal Investigator — Natera, Inc.
Locations (1):
- San Carlos, San Carlos, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kasi PM, Sawyer S, Guilford J, Munro M, Ellers S, Wulff J, Hook N, Krinshpun S, Koyen Malashevich A, Malhotra M, Rodriguez A, Moshkevich S, Grothey A, Kopetz S, Billings P, Aleshin A. BESPOKE study protocol: a multicentre, prospective observational study to evaluate the impact of circulating tumour DNA guided therapy on patients with colorectal cancer. BMJ Open. 2021 Sep 24;11(9):e047831. doi: 10.1136/bmjopen-2020-047831. PMID 34561256